CLINICAL TRIAL: NCT06381076
Title: Examining the Impact of High-protein Oral Supplement With Liposomal Curcumin on Inflammation Markers and Oxidative Stress in Adults Undergoing Hemodialysis.
Brief Title: High-protein Oral Supplement With Liposomal Curcumin in Adults Undergoing Hemodialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202400087
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease 5D

STUDY DESIGN:
Intervention Model Description: Randomized comparator-controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants will receive a 3-digit coded product that either contains 7 mls of liposomal curcumin or food colorant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will consume 38 g of high protein product with 7 mls of curcumin at the end of each dialysis session, 3 days a week for 8 weeks for a total of 24 treatments.
  Interventions: Drug: Liposomal curcumin
- Control (Placebo Comparator): Participants will consume 38 g of high protein product that contains an orange food colorant at the end of each dialysis session, 3 days a week for 8 weeks for a total of 24 treatments.
  Interventions: Drug: Food colorant

INTERVENTIONS:
Drug: Liposomal curcumin — participants will consume the product ad libitum for the 24 treatments.
  Other Names: Manna Liposomal Curcumin
  Arms: Intervention
Drug: Food colorant — participants will consume the product ad libitum for the 24 treatments as a placebo.
  Other Names: ChefMaster
  Arms: Control

SUMMARY:
A 12-week double-blind randomized control trial will be conducted among adults on hemodialysis (n=15) to determine the impact of liposomal curcumin in a high-protein product on inflammation markers and oxidative stress. Participants will be randomized via a computer-generator into either the control or intervention group. Participants in each group will be given a total of 38 g of a high protein product with or without 7 mls of liposomal curcumin for a total of 8 weeks. At baseline, weeks 8 and 12, participants will have blood sampled and complete a 3-day 24-hour recalls (2 non-dialysis days and 1 dialysis day) and a quality of life survey.

DETAILED DESCRIPTION:
This is a 12-week double-blind randomized controlled trial to evaluate the impact of liposomal curcumin in a high-protein product on inflammation markers for adults undergoing hemodialysis. CRP and oxidative stress will be assessed from monthly blood samples using Elisa kits. Quality of life will be measured using the standard 36-item kidney disease quality of life instrument. There will be a 2-month recruitment period prior to the start of the trial to ensure the potential participants are familiarized with the clinical trial. Eligible participants will sign the consent form to participate in the study. Once the expected number of participants has been reached, they will be randomized 1:1 using block randomization. Randomization will be done using a computer-generated program.

The intervention will take place over an 8-week period. Participants will have their blood drawn at the beginning of the study by the dialysis practitioner and start receiving the product on their next scheduled dialysis appointment. Participants will be receiving the product three times a week in accordance with their dialysis schedule (M-W-F or T-Th-S), for a total of 24 treatments. Blood will be collected at baseline, at the end of the study and a month after to assess any carryover effects. Additionally, participants will complete 3-day 24-hour recalls (2 non-dialysis days and 1 dialysis day), a spice-consumption survey, and a quality-of-life assessment at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* diagnosed with stage 5 CKD.
* receiving hemodialysis at least three months before the trial start date
* All participants can provide signed informed consent, have no dietary restrictions, no food allergies, nor chewing/swallowing difficulties.

Exclusion Criteria:

* Adults with CKD stages 1-4.
* Adults undergoing peritoneal dialysis.
* Pregnant and/or lactating for the duration of the study as confirmed by the dialysis medical staff.
* Use of other IP within 3 months of the initiation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
high-sensitivity C-reactive protein | 12 weeks or 84 days
  baseline to end line in the concentration of high-sensitivity C-reactive protein between the control and intervention group.

SECONDARY OUTCOMES:
Advanced glycation end products | 12 weeks or 84 days
  baseline to end line in the concentration of advanced glycation end products between the control and intervention group.
fatty acid byproduct - 4-hydroxynon-enal | 12 weeks or 84 days
  baseline to end line in the concentration of fatty acid byproduct - 4-hydroxynon-enal between the control and intervention group.
fatty acid byproduct - malondialdehyde | 12 weeks or 84 days
  baseline to end line in the concentration of fatty acid byproduct - malondialdehyde between the control and intervention group.
fatty acid byproduct - 8-F2 isoprostanes | 12 weeks or 84 days
  baseline to end line in the concentration of fatty acid byproduct - 8-F2 isoprostanes between the control and intervention group.
Klotho | 12 weeks or 84 days
  baseline to end line in the concentration of klotho between the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette M Andrade, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No